CLINICAL TRIAL: NCT00003229
Title: A Phase I-II Trial of Antigen-Pulsed Autologous Dendritic Cells for Induction of Anti-Tumor Immunity in Patients Completing Lymphadenectomy for Metastatic Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma Who Are Undergoing Surgery for Lymph Node and Tumor Removal
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066097; DUMC-719975; DUMC-0932-99-5R2; DUMC-759-99-5R2; UVA-HIC-7454; NCI-G98-1398
Record Dates: First submitted 1999-11-01; First posted 2004-08-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: gp100 antigen
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells and melanoma cells may make the body build an immune response and kill the tumor cells.

PURPOSE: Randomized phase I/II trial to study the effectiveness of vaccine therapy made from white blood cells and melanoma cells in treating patients with metastatic melanoma who are undergoing surgery for lymph node and tumor removal.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and toxicity of intravenous injections of autologous cultured dendritic cells pulsed with either gp100 and tyrosinase peptides or autologous melanoma tumor cell lysates in patients with metastatic melanoma. II. Determine whether treatment with melanoma tumor antigen pulsed autologous dendritic cells results in increased in vitro tumor specific cytotoxic T-cell responses. III. Determine whether this treatment can induce positive skin test responses to tumor antigens. IV. Evaluate the disease free and overall survival of these patients.

OUTLINE: This is a randomized, dose escalation study. Approximately 1-2 weeks following surgical lymphadenectomy, patients undergo leukapheresis to collect dendritic cells and are then divided into 3 groups. Group A consists of patients without adequate tumor for preparation of tumor lysate and who have tumors that express tyrosinase or gp100 with types HLA-A1, A2, or A3. Group B consists of the patients who have adequate tumor for lysate preparation but who do not type for HLA-A1, A2, or A3 (required for the peptide pulsed protocol). Group C are the patients with adequate tumor who are eligible for the peptide pulsed protocol. Group A patients receive autologous dendritic cells pulsed with appropriate peptide antigens. Group B patients are treated with autologous dendritic cells pulsed with autologous tumor cell lysates. Group C patients are randomized to receive dendritic cells pulsed with either peptide antigens or tumor lysate. All patients are administered intravenous active immunotherapy for 4 monthly intervals. The dose of the immunizations is escalated for each cohort of three patients that is accrued in each of the groups mentioned above. Each immunization at each dose level is followed by three days of interleukin-2 administered subcutaneously twice daily. Patients are followed at least 5 years for survival.

PROJECTED ACCRUAL: There will be 100 patients accrued in this study over 2 years. There will be 50, 20, and 30 patients in groups A, B, and C, respectively.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic melanoma involving cervical, axillary, inguinal, groin, or iliac lymph nodes All gross disease is resected at the time of surgical lymphadenectomy No distant metastases

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: ECOG 0-1 Life expectancy: At least 6 months Hematopoietic: Platelet count at least 100,000/mm3 Hemoglobin at least 8 g/dL Hepatic: Bilirubin no greater than 1.4 mg/dL AST or ALT no greater than 1.5 times normal No active hepatitis Renal: Creatinine no greater than 1.4 mg/dL Cardiovascular: No congestive heart failure, unstable angina, or current symptomatic arrhythmias Other: HIV negative No autoimmune diseases (e.g., lupus erythematosus, multiple sclerosis, or ankylosing spondylitis) No condition that would be considered as a contraindication for surgery Not pregnant or nursing Adequate contraception required for all fertile patients

PRIOR CONCURRENT THERAPY: At least 4 weeks since prior therapy for melanoma Biologic therapy: At least 3 months since prior interferon therapy Chemotherapy: No active immunosuppression due to prior chemotherapy Endocrine therapy: No active immunosuppression due to steroid therapy Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-07; Primary Completion 2000-04 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilliard F. Seigler, MD, Study Chair — Duke Cancer Institute
Locations (2):
- United States (2):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia